CLINICAL TRIAL: NCT06087692
Title: Efficacy of Video-Based Interactive Game Therapy in Interstitial Lung Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Melike Sarıtas Arslan, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PHD Thesis
Record Dates: First submitted 2023-10-06; First posted 2023-10-18 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Interstitial Lung Disease
Keywords: Video-based game therapy; Aerobic Exercise
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized-Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise (Other): Patients in the aerobic exercise group will be included a medium intensity (%40-60 of the maximum heart rate or 4-6 intensity according to the Modified Borg Scala) aerobic exercise program with a horizontal bicycle ergometer, 2 days a week for 8 weeks, lasting an average of 30 minutes, accompanied by a physiotherapist.
  Interventions: Other: Exercise
- Nintendo +aerobic exercise (Other): Nintendo group will be included a medium intensity (40-60% of the maximum heart rate or 4-6 intensity according to the Modified Borg scale) aerobic exercise program with a horizontal bicycle ergometer 2 days a week for 8 weeks, lasting an average of 30 minutes, accompanied by a physiotherapist, and then they will be included in ''Wii Fit'' exercise program an average of 30 minutes.
  Interventions: Other: Exercise
- Control (Other): Physical activity recommendation and respiratory exercises
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — -based game therapy applied in addition to aerobic exercise

SUMMARY:
Interstitial lung disease (ILD) is a heterogeneous group of diseases consisting of variable amounts of inflammation and fibrosis and a wide variety of acute and chronic pulmonary disorders affecting both the interstitium and lung parenchyma. The use of gamification elements in order to encourage changes in health behaviors such as physical activity appears as an entertaining option by increasing extrinsic motivation in sedentary individuals or in diseases where physical activity is targeted. The aim of this study is to investigate the effectiveness of Nintendo Wii applied in addition to aerobic exercise in patients with ILD on exercise capacity and peripheral muscle strength, symptoms, activity and participation with objective methods, based on evidence.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is a heterogeneous group of diseases consisting of variable amounts of inflammation and fibrosis and a wide variety of acute and chronic pulmonary disorders affecting both the interstitium and lung parenchyma. Many forms of ILD are progressive over time, associated with severely disabling symptoms and poor quality of life, yet medical treatment options are often limited. There are no specific pulmonary rehabilitation guidelines for this patient population, and standard programs are adapted on a patient basis. However, it is seen that the participation and attendance of patients in pulmonary rehabilitation programs is low, and the benefits obtained from the programs are gradually lost after completing the intensive rehabilitation process and breaking contact with the rehabilitation team. For these reasons, the guidelines emphasize the need to implement new strategies that can overcome limitations, and it is stated that there is a need for research and development of new program models that will make evidence-based pulmonary rehabilitation more accessible for patients. The use of gamification elements in order to encourage changes in health behaviors such as physical activity appears as an entertaining option by increasing extrinsic motivation in sedentary individuals or in diseases where physical activity is targeted. The aim of this study is to investigate the effectiveness of Nintendo Wii applied in addition to aerobic exercise in patients with ILD on exercise capacity and peripheral muscle strength, symptoms, activity and participation with objective methods, based on evidence.

Hypotheses:

H0: Video-based game therapy applied in addition to aerobic exercise in patients with ILD has has no effect on exercise capacity, quality of life and physical fitness level.

H1: Video-based game therapy applied in addition to aerobic exercise in patients with ILD increases exercise capacity, quality of life and physical fitness level.

Patients in the Nintendo group will be included a medium intensity (40-60% of the maximum heart rate or 4-6 intensity according to the Modified Borg scale) aerobic exercise program with a horizontal bicycle ergometer 2 days a week for 8 weeks, lasting an average of 30 minutes, accompanied by a physiotherapist, and then they will be included in ''Wii Fit'' exercise program an average of 30 minutes. Patients in the aerobic exercise group will be included a medium intensity (%40-60 of the maximum heart rate or 4-6 intensity according to the Modified Borg Scala) aerobic exercise program with a horizontal bicycle ergometer, 2 days a week for 8 weeks, lasting an average of 30 minutes, accompanied by a physiotherapist. After eight weeks, all assessments will be repeated.

As a result of this study, the contribution of video-based interactive game therapy to exercise capacity, peripheral muscle strength, physical activity level, symptoms, activity and participation levels in patients with ILD will be determined and compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ILD (Interstitial lung disease) by a chest diseases specialist, aged between 40-65 years, and have been under follow-up for at least 6 months according to the current ATS/ERS guidelines.
* Clinically stable, with no exacerbations or infections.
* Able to walk, with no visual or auditory impairments.
* Patients with cognitive abilities sufficient to understand commands.

Exclusion Criteria:

Orthopedic and neurological problems that could hinder exercise training.

* Changes in medical treatment during the study.
* Unstable cardiac diseases.
* Insufficient cooperation.
* Diagnosed visual, auditory, vestibular, or neurological problems that could affect balance.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | through study completion, an average of 1 year
  6 minute walk test:Used to determine submaximal functional exercise capacity. Patients are asked to walk as far as possible in a 30-meter straight corridor at their own walking pace for six minutes. The patient rests in a sitting position for 10 minutes in the corridor before starting the test. Oxygen saturation, heart rate, blood pressure, dyspnea, and leg fatigue scores are recorded before and after the test. The distance walked in six minutes is recorded.
Incremental Shuttle Walk Test | through study completion, an average of 1 year
  Incremental Shuttle Walk Test (ISWT): Used to determine functional exercise capacity. Patients walk around a cassette with signals previously recorded at a rate of 0.17 m/s, which increases every minute, starting at a pace of 10 meters per minute. The test consists of a maximum of 12 stages. The test is terminated if the patient cannot complete it within the allowed time (if the patient is more than 0.5 meters away from the signal cone when the signal sounds) or if the patient reaches 85% of the predicted maximum heart rate calculated according to the formula [210 - (0.65 x age)]. Oxygen saturation, heart rate, blood pressure, dyspnea, and leg fatigue scores are recorded before and after the test. The walking distance is recorded.
Endurance Shuttle Walk Test | through study completion, an average of 1 year
  Endurance Shuttle Walk Test (ESWT): Endurance capacity is determined using ESWT. The walking speed (workload) to be used in ESWT will be calculated as 85% of the maximum sustainable speed obtained from ISWT. Patients are asked to warm up by walking at a slower pace for two minutes and then to walk at a steady pace. The test is terminated if the patient feels too breathless to continue walking, becomes fatigued, or completes the 20-minute test duration. Oxygen saturation, heart rate, blood pressure, dyspnea, and leg fatigue scores are recorded before and after the test. The walking time is recorded in seconds.

SECONDARY OUTCOMES:
Respiratory Muscle Strength | through study completion, an average of 1 year
  Measurement of respiratory muscle strength will be performed using an electronic mouth pressure measurement device, the "MicroRPM" brand (Micro Medical; UK), in accordance with ATS and ERS criteria.
Muscle strength | through study completion, an average of 1 year
  Quadriceps Function Assessment;Quadriceps muscle strength will be evaluated using a hand-held dynamometer (J-Tech CommanderTM Muscle Tester, USA) by performing maximal voluntary isometric contractions (break test).
Dyspnea | through study completion, an average of 1 year
  The Modified Medical Research Council Scale is used to assess the level of dyspnea experienced in daily life.The Medical Research Council (MRC) Scale for Muscle Strength is a commonly used scale for assessing muscle strength from Grade 4 (normal) to Grade 0 (no visible contraction).
Fatigue | through study completion, an average of 1 year
  A 9-item Fatigue Severity Scale is created by selecting fatigue-related characteristics. Each question is rated on a scale of 1-7, with 1 indicating no effect and 7 indicating a high impact. The total score is calculated as the sum or average of all responses.
The Saint George Respiratory Questionnaire | through study completion, an average of 1 year
  The Saint George Respiratory Questionnaire (SGRQ) is used to assess health-related quality of life. It consists of 50 questions and three subscales: symptoms, activity, and impact.Scores range from 0 to 100, with higher scores indicating more limitations.
Daily Life Activities: | through study completion, an average of 1 year
  The London Chest Activity of Daily Living Scale (LCADL) is used to assess daily life activities and their impact on breathlessness. The scale has 4 subgroups; self-care (4 question), about home (six question), physical activity (2 question) and leisure time (3 question). The minimum score is 0 and maximum score is 75. Higher scores indicate worse conditions.
International Physical Activity Questionnaire (Short Form) | through study completion, an average of 1 year
  This questionnaire is used to determine the level of physical activity.
  1. Inactive-No activity is reported OR
     • Some activity is reported but not enough to meet Categories 2 or 3.
  2. Minimally Active Any one of the following 3 criteria
     * 3 or more days of vigorous activity of at least 20 minutes per day OR
     * 5 or more days of moderate-intensity activity or walking of at least 30 minutes per day OR
     * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-min/week.
  3. active Any one of the following 2 criteria
     * Vigorous-intensity activity on at least 3 days and accumulating at least 1500 METminutes/week OR
     * 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET-minutes/week
Leicester Cough Questionnaire | through study completion, an average of 1 year
  Leicester Cough Questionnaire (LCQ) is an English-born self-reporting quality of life measure of chronic coug. It consists of 19 items with a 7 point likert response scale (range from 1 to 7). Each item is developed to assess symptoms during cough and impact of cough on three main domains: physical, psychological and social. Scores are calculated as a mean of each domain and the total score is calculated by adding every domain score. It generally takes about 5 minutes to be completed and it is designed for adults.The total severity score ranges from 3 to 21, with a lower score indicating greater impairment of health status due to cough.
Global rating of change (GRC) | through study completion, an average of 1 year
  Global rating of change (GRC): Patient satisfaction was assessed by GRC at the end of the study. Global rating of change (GRC) scales are designed to quantify a patient's improvement or deterioration over time, usually either to determine the effect of an intervention or to chart the clinical course of a condition (21). The responses for the GRC were "much better"; "slightly better"; "stayed the same"; "slightly worse" or "much worse".

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yıldız Özer, Prof., Study Director — Marmara University
Locations (1):
- İstanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holland AE, Hill CJ, Conron M, Munro P, McDonald CF. Short term improvement in exercise capacity and symptoms following exercise training in interstitial lung disease. Thorax. 2008 Jun;63(6):549-54. doi: 10.1136/thx.2007.088070. Epub 2008 Feb 1. PMID 18245143
- [Derived] Arslan MS, Ozer AY, Bingol Z, Okumus G. Effectiveness of Active Video Games as a Training Tool in Patients With Interstitial Lung Disease: A Randomised Controlled Trial. Respirology. 2025 Dec 4. doi: 10.1002/resp.70166. Online ahead of print. PMID 41344887